CLINICAL TRIAL: NCT05904067
Title: Institute of Hematology & Blood Diseases Hospital
Brief Title: A Study to Evaluate the Safety and Efficacy of COVID-19 Convalescent Plasma (CCP) Transfusion to Prevent COVID-19 in Adult Recipients Following Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCP-COVID-19-HSCT-2023
Record Dates: First submitted 2023-06-13; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: COVID-19; Hematopoietic Stem Cell Transplantation
Keywords: COVID-19 Convalescent Plasma; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recipient of COVID-19 Convalescent Plasma (CCP) Transfusion (Experimental): Transfusion of COVID-19 convalescent plasma to participants The experimental group (CCP group): 200 ml of CCP at +14 days, +28 days, +2 months, and +3 months following hematopoietic stem cells transplantation.
  Interventions: Biological: COVID Convalescent Plasma
- Recipient without COVID-19 Convalescent Plasma (CCP) Transfusion (No Intervention): Control group (supportive therapy): patients were routinely given oral ursodeoxycholic acid for +14 days after transplantation.

INTERVENTIONS:
Biological: COVID Convalescent Plasma — 200 ml of COVID Convalescent Plasma at +14 days, +28 days, +2 months, and +3 months following hematopoietic stem cells transplantation.
  Other Names: CCP, COVID-19 Convalescent Plasma
  Arms: Recipient of COVID-19 Convalescent Plasma (CCP) Transfusion

SUMMARY:
The study is to evaluate the safety and efficacy of COVID-19 convalescent plasma (CCP) transfusion to prevent COVID-19 in adult recipients following hematopoietic stem cell transplantation.

72 patients will be randomized in a 1:1 ratio to receive either CCR (36 patients) or not (36 patients). Patients in the CCP group will receive 200 ml of CCP at +14 days, +28 days, +2 months, and +3 months following hematopoietic stem cell transplantation. Patients in the control group would be routinely given oral ursodeoxycholic acid for +14 days after transplantation.

The primary goal of the study is to evaluate the safety of CCP and the incidence of COVID-19 infection within +28 days after the last infusion of CCP.

ELIGIBILITY:
Inclusion Criteria:

1. receive hematopoietic stem cell transplantation
2. Be ≥ 16 years of age on the day of enrollment.
3. Understand the study procedures, alternative treatment available, and risks involved with the study, and voluntarily agree to participate by giving written informed consent.

Exclusion Criteria:

1. Positive serological response to known HIV or active hepatitis C virus.
2. Patients with mental illness or other conditions that do not meet the requirements of research treatment and monitoring.
3. Unable or unwilling to sign consent form.
4. Patients with other special conditions assessed as unqualified by the researchers.
5. Patients suffered COVID-19 infection between day 0 and infusion of CCP after transplantation.

Drop-out and Withdrawal Criteria

1. Failure of engraftment within 30 days of transplantation;
2. Patients who are not compliant with the requirements of the study and fail to follow the study plan.
3. Patients receiving prophylaxis for COVID-19 infection by methods other than this protocol during the trial.
4. A patient may withdraw from the study if he/she does not wish to continue participating in the study, and the date and reason for withdrawal shall be recorded. The investigator may also decide to discontinue a patient from the clinical study if there is an unacceptable risk.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-06-10 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the prevalence of new COVID infection | 1 year
  within +28 days after the last infusion of CCP

SECONDARY OUTCOMES:
To evaluate the incidence of severe COVID-19 | 1 year
  within +28 days after the last infusion of CCP
To evaluate the survival rate of COVID-19 infection | 1 year
  within 30 days after COVID-19 infection within +28 days after last CCP infusion
To evaluate the overall survival | 1 year
  at 1 year after transplantation.
To evaluate the tolerance of CCP infusion | 1 year
  at 1 year after transplantation.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, None Selected, China

REFERENCES:
- [Derived] Cao Y, Li Q, Guo W, Xu M, Fang K, Wang F, Zhang R, Li L, Wei J, Liu Z, Liang C, Zhai W, Ma Q, Chen X, Cao W, Yang D, He Y, Pang A, Feng S, Han M, Sun J, Jiang E. Convalescent plasma therapy for COVID-19 prophylaxis in adults early post-hematopoietic stem cell transplantation: one-year outcomes from a randomized controlled trial. Front Immunol. 2025 Nov 28;16:1626775. doi: 10.3389/fimmu.2025.1626775. eCollection 2025. PMID 41394817